CLINICAL TRIAL: NCT04168879
Title: Efficacy of Suprazygomatic Approach of Sphenopalatine Ganglion Block for Nasal Surery
Brief Title: Sphenopalatine Ganglion Block for Nasal Surery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Collaborators: saeid metwaly abouelyazid elsawy (Unknown)
Responsible Party: Principal Investigator, Rasha Hamed, lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ACCA
Record Dates: First submitted 2019-11-16; First posted 2019-11-19 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Emergence Agitation
MeSH Terms: conditions — Emergence Delirium | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bupivacaine group (Active Comparator)
  Interventions: Drug: Bupivacaine 0.5% Preservative-Free Injectable Solution
- saline group (Placebo Comparator)
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Bupivacaine 0.5% Preservative-Free Injectable Solution — 1.5 ml of Bupivacaine 0.5% Preservative-Free Injectable Solution used to block the sphenopalatine ganglion by ultrasound guided suprazygomatic approach
  Arms: bupivacaine group
Drug: normal saline — 1.5 ml of normal saline is delivered to the sphenopalatine ganglion by ultrasound guided suprazygomatic approach
  Arms: saline group

SUMMARY:
nasal surgery carries many perioperative challenges, intraoperative bleeing and its effect on surgical field i the main intraoperative concern an postoperative agitation and its serious complications is the main postoperative challenge.

ELIGIBILITY:
Inclusion Criteria:

* patient written consent
* elective surgery
* age 18 - 55 year old

Exclusion Criteria:

* patient refusal
* emergency surgery

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Postoperative emergence agitation | 2 hour
  ramsy hunt sedation agitation score used during emergence from anesthesia

SECONDARY OUTCOMES:
postoperative opioid consumption | 24 hour
  total amount of opioid analgesia in first 24 hours postoperative
surgical field quality | 2 hours
  Boezaart score was be used
consumed inhalational anesthesia | 2 hours
  mean anesthesia MAC intraoperative
postoperative pain | 2 hours
  using VAS ; scale from 0 to 10 . where 0 is no pain and 10 is worst pain

OTHER OUTCOMES:
intraoperative bleeding | 2 hours
  suction and weight of surgical gauze used was measured and calculated

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamed R, Gamal L, Elsawy S, Baker MA, Abbas YH. Efficacy of ultrasound guided sphenopalatine ganglion block in management of emergence agitation after sinoscopic nasal surgery: a randomized double-blind controlled study. Anaesth Crit Care Pain Med. 2024 Dec;43(6):101429. doi: 10.1016/j.accpm.2024.101429. Epub 2024 Oct 2. PMID 39366653